CLINICAL TRIAL: NCT07048951
Title: Episodes of (Dis)Connected Consciousness Among Patients Who Survived a Critical Illness
Brief Title: Episodes of (Dis)Connected Consciousness in ICU Survivors
Acronym: CONSCIOUS-ICU
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-254
Record Dates: First submitted 2025-04-07; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-12

CONDITIONS: Consciousness; Near Death Experience; ICU; Critical Illness
Keywords: near-death experience; out-of-body experience
MeSH Terms: conditions — Death; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survivors of prolonged ICU (≥7days) stay with episode(s) of pharmacological/non-pharmacological coma
  Interventions: Diagnostic Test: The Near-Death Experience Content (NDE-C) scale; Other: Threat perception measure; Other: Interview about the participant's memories of the ICU

INTERVENTIONS:
Diagnostic Test: The Near-Death Experience Content (NDE-C) scale — Questionnaire to detect occurence of NDE. A NDE is identified if score > or = 27/80
Other: Threat perception measure — 7 items scale investigating the participant's psychological vulnerability during their stay at the ICU
Other: Interview about the participant's memories of the ICU — Participants will be asked to describe any dream, hallucination, or any other unusual experience they can recall from their stay at the ICU.
  Additionally, the participants will be asked to describe any memory they have of the environment of the ICU, such as the appearance of the room, medical staff, family visiting, noises, etc.

SUMMARY:
This single-center observational study aims to describe the incidence of episodes of connected consciousness and disconnected consciousness (including near-death experience (NDE) and out-of-body experiences) in patients who survived a prolonged stay of at least 7 days in the intensive care unit (ICU) and who had at least one episode of pharmacological or non-pharmacological coma. The investigators are also investigating the risk factors related to these episodes of consciousness. A follow-up at six months aims to explore the long-term psychological implications of these episodes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who survived a ≥7 days stay in the intensive care unit
* Experienced a pharmacological or non-pharmacological episode of loss of consciousness
* French speaking

Exclusion Criteria:

* Refusal
* Chronic disorder of consciousness
* Confusion or delirium
* Deafness
* Blindness
* Aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Detection of potential episodes of disconnected consciousness | Within the week following discharge from the ICU (max 7 days after)
  Near-death experience (using the Near-Death Experience Content scale, min-max: 0-80, with ≥27/80 indicating the presence of a NDE); dream
Detection of potential episodes of connected consciousness | Within the week following discharge from the ICU (max 7 days after)
  Explicit recall of environmental/external stimuli in the ICU

SECONDARY OUTCOMES:
Risk factors | Within the week following discharge from the ICU (max 7 days after)
  (Neuro)physiological marker
Psychological vulnerability during the stay at the ICU | Within the week following discharge from the ICU (max 7 days after)
  Using the Threat Perception Measure, a scale that contains 7 items related to feelings and anxieties perceived by the patient, each scored from 1 to 4, ranging from 1 "Not at all", 2 "A little", 3 "Moderately", and 4 "Extremely", as well as a "don 't remember" category. Min-max: 7-28, with higher scores indicating a higher level of perceived threat
Psychological impact of the stay at the ICU | At a 6 month follow-up after discharge from the ICU
  Any patient who stayed at least 7 days at the ICU is invited to a 6 month follow-up during which they will be presented Hospital Anxiety and Depression Scale (HADS, min-max: 0-42, with higher scores indicating a worse outcome, i.e., more severe symptoms of anxiety or depression), to assess anxiety and depression as well as the Post-Traumatic Stress Assessment Questionnaire (IES-R, min-max: 0-88, with higher scores indicating a worse outcome, i.e., more severe post-traumatic stress symptoms).
  The investigators will be asking two additional questions to investigate a possible impact on the patient's beliefs.
  * Question 1: "Since your stay in intensive care, have your beliefs/opinions changed regarding death?".
  * Question 2: "Has your stay in intensive care modified your fear of health care institutions?

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Liège, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No